CLINICAL TRIAL: NCT05594797
Title: A Phase Ⅱ Clinical Study Evaluating the Efficacy and Safety of Human BCMA Targeted T Cells Injection Therapy for Relapsed/Refractory Multiple Myeloma
Brief Title: Human BCMA Targeted T Cells Injection（BCMA CAR-T）for Subjects With R/R MM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Changzheng Hospital (Other); First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-MM01-Ⅱ
Record Dates: First submitted 2022-10-18; First posted 2022-10-26 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: BCMA; CAR-T; Relapsed/Refractory; Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Human BCMA Targeted T Cells Injection (Experimental): Single administration：6.0×10^6 CAR+T/kg
  Interventions: Drug: Human BCMA Targeted T Cells Injection

INTERVENTIONS:
Drug: Human BCMA Targeted T Cells Injection — A single dose of predetermined level CAR-positive T cells will be infused.
  Other Names: BCMA CAR-T

SUMMARY:
A Phase Ⅱ Clinical Study Evaluating the Efficacy and Safety of Human BCMA Targeted T Cells Injection（BCMA CAR-T） Therapy for R/R MM.

Patients will be given a conditioning chemotherapy regimen of fludarabine and cyclophosphamide followed by a single infusion of BCMA CAR+ T cells.

DETAILED DESCRIPTION:
Participants with relapsed/refractory multiple myeloma can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, Electrocardiograph, Computedtomography （CT）/Magnetic Resonance Imaging(MRI)/Positron Emission Tomography（PET）, and blood draws. Participants receive chemotherapy prior to the infusion of BCMA CAR+ T cells. After the infusion, participants will be followed for side effects and effect of BCMA CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:Subjects must meet all of the following criteria to be enrolled:

* Subjects volunteer to participate in clinical trails, understand and inform the trials and sign informed consent form, be willing to complete all the trial procedures;
* 18 to 75 years old (including cut-off value)，gender is not limited;
* Expected survival > 12 weeks;
* Previously diagnosed as multiple myeloma by the International Myeloma Working Group（IMWG） updated criteria;
* One of the following indicators is satisfied:

  1. Serum M protein ≥ 5 g/L;
  2. Urine M protein ≥ 200 mg/24h;
  3. Affected serum free light chain ≥ 100 mg/L and Serum free light chain ratio is abnormal ;
* Patients with relapsed/refractory multiple myeloma, satisfying:

  1. Patients have received at least 3 prior MM treatment regimens containing at least one proteasome inhibitor and one immunomodulator;
  2. Progress is documented within 12 months of the most recent antimyeloma treatment, or efficacy assessment does not reach minimal response(MR) or above or progression within 60 days of the most recent antimyeloma treatment;
* ECOG score 0-2;
* Autologous hematopoietic stem cell transplantation is not possible or relapses after autologous hematopoietic stem cell transplantation, but requires further treatment at the investigator's discretion；
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Creatinine clearance rate (estimated by CockcroftGault formula)≥40mL/min;
  2. Total bilirubin≤2×ULN; Alanine aminotransferase (ALT) ≤2.5×ULN and aspartate aminotransferase (AST)≤2.5×ULN;
  3. Left ventricular ejection fraction >50%;
  4. Baseline peripheral oxygen saturation>95%;
* The venous access required for collection can be established, no contraindications to leukocyte collection, and leukepheresis can be carried according to the judgement of investigators, satisfying hemoglobin≥70g/L,platelets ≥50×10^9 / L, neutrophils ≥1.0×10^9/L.

Exclusion Criteria:Any one of the following conditions cannot be selected as a subject：

* Subjects have a history of central nervous system (CNS) diseases such as seizures, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, psychosis; known or history of active central nervous system (CNS) involvement or presentation of multiple myeloma meninge/meningeal involvement;
* Subjects with plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome, or primary light chain amyloidosis;
* Accompanied by other uncontrolled malignancies, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection and thyroid cancer after radical resection ;
* Any uncontrollable active infection, including but not limited to active tuberculosis; fungal, bacterial, viral, or other infections that are uncontrollable or require systemic intravenous therapy are present or suspected within 14 days prior to enrollment;
* Subjects with positive Hepatitis B surface antigen(HBsAg) or Hepatitis B core antibody (HBcAb) and hepatitis B virus (HBV) DNA titers higher than the lower limit of the normal range of the investigative site); Hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; Human Immunodeficiency Viral (HIV) antibody positive; syphilis positive;
* Any uncontrolled systemic diseases, including but not limited to unstable angina pectoris, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ Ⅲ), uncontrolled diabetes mellitus (glycosylated hemoglobin HbAlc >8% at screening)，severe arrhythmia, liver, kidney, or metabolic diseases that are poorly controlled by medications;
* Subjects who have a history of pacemaker and brain pacemaker implantation;
* Subjects who have received CAR-T treatment or other genetically modified cell therapies, as well as other BCMA-targeting drugs;
* Subjects with any hematopoietic stem cell transplant performed within the first two months of screening, or any immunosuppressive therapy due to graft-versus-host disease performed during the screening period;
* Subjects who were receiving systemic steroid treatment within 14 days before the screening period and who were judged by the investigator to require long-term use of systemic steroid therapy during treatment (except inhalation or topical use); or subjects who received any systemic anti-tumor therapy ( except for local anti-tumor therapy) ;
* Subjects who have received live attenuated vaccine within 4 weeks prior to apheresis;
* In the past two years, the terminal organ was damaged due to autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), or the systemic use of immunosuppressive or other systemic disease control drugs was required;
* Pregnant or lactating woman, or planned pregnancy during treatment or within 1 year after treatment, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion; except participants of childbearing age are willing to use a very effective and reliable method of contraception for 1 year after study treatment;
* Subjects who have a disease that affects the signing of written informed consent or who are unable to comply with research procedures; or who are unwilling or unable to comply with research requirements;
* Subjects who have had severe immediate hypersensitivity reactions to any drugs used in this research;
* Subjects who are considered unsuitable to participate in this trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) at 3 months post infusion as evaluated by the Independent Review Committee | 3 months post infusion
  ORR at 3 months post infusion as evaluated by the Independent Review Committee (IRC) includes stringent complete response (sCR), complete response (CR), very good partial response (VGPR), and partial response (PR).

SECONDARY OUTCOMES:
Duration of remission (DOR) after administration | 2~3 years post infusion
  DOR refers to the time from the first assessment of the tumor for complete response and above efficacy to the first assessment of disease progression or death of any cause;
Progression-free Survival (PFS) after administration | 2~3 years post infusion
  PFS refers to the time from the start of cell infusion to the first assessment of tumor progression or death from any cause;
Overall Survival (OS) after administration | 2~3 years post infusion
  OS refers to the time from cell infusion to death due to any cause;
Objective Response Rate (ORR) at 3 months post infusion as evaluated by the Investigator | 3 months post infusion
  ORR at 3 months post infusion as evaluated by the Investigator;
Objective Response Rate (ORR) at 6 months post infusion as evaluated by the Independent Review Committee | 6 months post infusion
  ORR at 6 months post infusion as evaluated by the Independent Review Committee (IRC)；
Percentage of Subjects With Negative Minimal Residual Disease (MRD) | 2~3 years post infusion
  MRD negative rate is defined as the proportion of subjects who achieve MRD negative status;
Duration of Subjects With Negative Minimal Residual Disease (MRD) | 2~3 years post infusion
  MRD duration will calculated among MRD negative responders fom the date of initial MRD negative to the date of first documented evidence of MRD positive, as defined in the International Myeloma Working Group（IMWG） criteria (2016);
Number of Subjects with Adverse Events | 2~3 years post infusion
  Adverse event is any untoward medical event that occurs in a subject administered an investigational drug.
Change from Baseline in Perform Status as Measured by Eastern Cooperative Oncology Group（ECOG）Score（0-2） | 2~3 years post infusion
  Eastern Cooperative Oncology Group（ECOG） Performance Status Score（0-2） will be assessed by the inverstigator at baseline and the respective time point, higher scores mean a worse performance status.
The occurrence rate of adverse events grade ≥ 3 assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. | 2~3 years post infusion
  Safety Indicators
Change in body weight over time after reinfusion | 2~3 years post infusion
  Safety Indicators
Pharmacokinetic indicators:Maximum CAR level inperipheral blood or bone marrow (Cmax) | 2~3 years post infusion
  The highest concentration of Human BCMA Targeted T Cells Injection amplified in peripheral blood or bone marrow after infusion (Cmax) ；
Pharmacokinetic indicators: Time to peak CAR level in blood or bone marrow (Tmax) | 2~3 years post infusion
  The time to reach the highest concentration of Human BCMA Targeted T Cells Injection in peripheral blood or bone marrow after infusion (Tmax) ；
Pharmacokinetic indicators: 28-day Area under the curve of the CAR level in blood or bone marrow (AUC0-28d) | 2~3 years post infusion
  The 28-day area under the curve of Human BCMA Targeted T Cells Injection in peripheral blood or bone marrow after infusion（AUC0-28d）；
Pharmacodynamic indicators: the concentration level of soluble BCMA (sBCMA) in peripheral blood | 2~3 years post infusion
  The concentration level of soluble BCMA (sBCMA) in peripheral blood at various time points after infusion of Human BCMA Targeted T Cells Injection；
Pharmacodynamic indicators: the concentration level of CAR-T cell-related serum cytokines such as C-Reactive Protein（CRP） in peripheral blood； | 2~3 years post infusion
  Effectiveness Metrics
Pharmacodynamic indicators: the concentration level of CAR-T cell-related serum cytokines such as Interleukin-6（IL-6）, IL-2, IL-10, Tumor Necrosis Factor （TNF-α），Interferon-γ（IFN-γ）in peripheral blood； | 2~3 years post infusion
  Effectiveness Metrics
Immunogenicity: Anti-drug antibody(ADA) positive ratio | 2~3 years post infusion
  Immunogenicity study evaluated the immune responses to anti-BCMA scFV including the detection of anti-scFV antibodies；
Immunogenicity: Neutralizing Antibody(Nab) positive ratio | 2~3 years post infusion
  Immunogenicity study evaluated the immune responses to anti-BCMA scFV including the detection of neutralizing antibodies (NAbs) against scFV.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Ph.D., Principal Investigator — Shanghai Changzheng Hospital; Songfu Jiang, Professor, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (2):
- China (2):
  - Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No